CLINICAL TRIAL: NCT05241522
Title: A Phase 1, Open-Label Study to Investigate the Dosimetry of Tc-99m-Tilmanocept Following a Single Intravenous Dose Administration in Women and Men Suspected of Diabetic Nephropathy.
Brief Title: Dosimetry of Tc-99m-Tilmanocept
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Carl Hoh, Prof-hcomp - Radiology, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DK127201-02
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tilmanocept Dose - 0.050 mg (Active Comparator)
  Interventions: Diagnostic Test: Tc-99m-Tilmanocept
- Tilmanocept Dose - 0.20 mg (Active Comparator)
  Interventions: Diagnostic Test: Tc-99m-Tilmanocept
- Tilmanocept Dose - 0.40 mg (Active Comparator)
  Interventions: Diagnostic Test: Tc-99m-Tilmanocept

INTERVENTIONS:
Diagnostic Test: Tc-99m-Tilmanocept — Administration of 3 different doses of Tc-99m-Tilmanocept prior to SPECT-CT imaging of the kidney in order to determine the safety and efficacy of tilmanocept imaging for differentiating diabetic kidney disease from other causes of kidney disease.

SUMMARY:
This proposal will use kidney SPECT/CT of Tc-99m-tilmanocept to evaluate the mesangial changes seen in diabetics across the spectrum of kidney disease as well as persons with hypertensive kidney disease, the next most common cause of kidney disease in patients with diabetes. We aim to demonstrate that these different disease types and stages can be differentiated with Tc-99m-tilmanocept SPECT/CT and can thus be used for future trials evaluating early diagnosis and treatment of diabetic nephropathy.

DETAILED DESCRIPTION:
In this open-label, non-randomized, single center study all subjects will receive IV administration of one of 3 tilmanocept mass doses: 0.050 mg, 0.20 mg, and 0.40 mg all radiolabeled with 10 mCi technetium Tc-99m. A total of 120 subjects will be enrolled in this study. 30 subjects in each group will be recruited (total 120). Within each study group, 10 subjects will receive one of the 3 doses mentioned above.

We will start with the lowest molar dose (0.050 mg tilmanocept). Within this dose level we will first study ten patients with normal renal function (Group 1), followed by ten Group 2 patients, ten Group 3 patients, and ten Group 4 patients. This sequence will be repeated at the middle dose level (0.20 mg tilmanocept), and finally at the highest dose (0.40 mg tilmanocept).

Group 1 No evidence of CKD: Participants in this group must have an eGFR >60/ml/min/1.73m2 and a urine albumin to creatinine ratio of <30 mg/g at the time of enrollment.

Group 2 Stage 3a CKD: Participants in this must an eGFR of 45 - 60 /ml/min/1.73m2 Group 3 Stage 3b CKD: Participants in this must an eGFR of 30 - <45 /ml/min/1.73m2 Group 4 Stage 4 CKD: Participants in this must an eGFR of 15 - <30 /ml/min/1.73m2 Participants within each group will be recruited in a 1:1 fashion, of diabetic vs non diabetic, such that within each group, there will be 30 participants, 15 with diabetes and 15 without diabetes. Diabetes will be defined as a history of a hemoglobin A1c >6.5 and an on at least 1 anti-hyperglycemic agent.

In this study subjects will be asked to come in for 4 visits: A screening visit for initial determination of eligibility and evaluation of clinical status (Visit 1), a baseline visit, Day 1 (Visit 2), on the day of tilmanocept administration and imaging, a visit one day after tilmanocept administration Day 2 (Visit 3), and a 5 -7 day safety follow-up (Visit 4).

The IV administration will be performed Nuclear Medicine clinic at UCSD Medical Center, Hillcrest by an onsite Certified Nuclear Medicine Technologist or Nuclear Medicine Physician. All other visits will be done at UCSD Medical Center, La Jolla.

All the procedures listed below are experimental and considered part of the research study.

Screening Visit 1 (Day -29 to Day 0) This visit may be conducted over the phone followed by an in-person research visit for blood draw and urine collection.

* Preliminary review of inclusion and exclusion criteria (PHS Human Studies & Clinical Trial Info for complete list)
* Obtain signed informed consent for study participation.
* Allocation of unique subject number; this number will be used to document the subject data in the case report forms (CRFs) and enrollment log
* Demography - date of birth, gender, race
* Medical/surgical history- Medical/Surgical history will be obtained on all study subjects. All relevant prior medical and surgical conditions will be recorded in the eCRFs. Documented medical conditions will also note the month and year of onset if the condition is still active
* Concomitant Medications (within 30 days before injection)
* Vital signs (body temperature, heart rate, blood pressure, and will be collected from the SOC visit.
* Any clinically significant abnormal findings will be noted on the subject's medical history
* Clinical laboratory tests - study subjects will have blood obtained for hematology, chemistry and serology (HBsAg, HCV Ab, HIV)
* Urine collection for routine urinalysis and for pregnancy testing for women of child-bearing potential. Females of child-bearing potential are defined as women that are not surgically sterile (hysterectomy or bilateral oophorectomy) nor postmenopausal for at least 1 year prior to screening. Women who are not of childbearing potential will not require a pregnancy test
* 24-hour urine collection for estimate of 24 hour urine creatinine clearance. Visit 2 (Prior to Tc-99m-Tilmanocept Administration) All subjects will be assessed for adverse events in an ongoing manner from the day of injection through the end of participation. The following procedures will be completed on the day of injection prior to the administration of Tc-99m-tilmanocept: a urine pregnancy test for women of child-bearing potential, assessment of adverse events, concomitant medication review, ECG within 15 minutes prior to administration of Tc-99m- tilmanocept, vital signs after at least 1 minute in a resting position (heart rate, blood pressure,respiratory rate and weight) within 15 minutes prior to administration of Tc-99m-tilmanocept, IV catheter placement (preferably the left and right antecubital veins),and pre-Dose blood draw for chemistry and hematology. In addition, a physical examination will be done. This will include examination of general appearance, skin, eyes, ears, nose, throat, head and neck (including thyroid), lungs, heart, abdomen, lymph nodes, musculoskeletal, and nervous system. Any clinically relevant finding is to be documented as baseline finding.

Lymphoseek radiolabeling kits will be purchased for Cardinal Health (see letter in the PHS Human Studies & Clinical Trials Form) and radiolabeled in the PET Production Facility in the UCSD Moores Cancer Center.

Intra-venous administration of Tc-99m-tilmanocept will be at study time 00:00. Subjects will have a 20-22- gauge intra-venous catheter placed in the antecubital vein. An intravenous T-connector extension (Medex MX453L T Conn w/MLL) will be used to allow a quantitative injection of the radiopharmaceutical with no residual trapping in the IV setup (Figure 1). The filled syringe will be connected to the catheter for a slow push (5 to 10 secs) injection. At the completion of the injection, a 10-cc sterile normal saline flush will be administered.

Dynamic planar imaging:

The subject imaging protocol is in Figure 2. The subject will be placed in the dual-headed SPECT/CT gamma camera gantry for simultaneous anterior and posterior planar imaging. The patient will be positioned so that the imaging field of the anterior and posterior camera heads cover the left ventricular cavity of the heart, all of the liver, and both the kidneys. The dynamic imaging study will start at the same time as the Tc-99m-tilmanocept injection (370 MBq,10 mCi). The dynamic study will consist of a set of planar images (anterior and posterior views) and will last for a total of 30 minutes. This acquisition will consist of:

1. 2 sec/frame x 30 frames, then
2. 10 sec/frame x 174 frames (ending at 30 minutes).
3. Blood samples (5 cc) (5±0.5, 15±1.5 & 30±3 minutes post-injection) with pre-sample discard (3 cc) will be obtained from the IV line (after removal of the T-connector).

Pre- & post-urination planar images (approximately 5 minutes each) Immediately after the dynamic imaging study, 5-minute (anterior & posterior) planar images of the urinary bladder will be acquired. Upon completion of the bladder images, the patient will urinate into a pre-weighed collection jar. This can occur within 40 minutes post-injection. After urination, the patient will be repositioned in the SPECT/CT scanner for a set (anterior & posterior) post-urination images of the bladder.

Heart/liver/kidney spect (approximately 30 minutes):

This portion of the imaging will be performed on a dual headed SPECT/CT scintigraphic camera fitted with LEAP collimators. Sixty-four 1-minute projections will be acquired with a 10% window centered at 140 keV, and a 128 x 128 image matrix.

Non-imaging procedures:

* ECG (completed before vital signs) within 15 minutes prior to Tilmanocept administration and at 30 minutes post-injection. (up to a total of 2 times at this visit)
* Vital signs after at least 1 minute in a resting position (heart rate, blood pressure, and respiratory rate) at 5 minutes, 15 minutes, 30 minutes, 60 minutes and 90 minutes. (up to a total of 6 times at this visit)
* Concomitant medication review.
* Assessment and review of adverse events.

Visit 3 (One Day after Tilmanocept Administration) & Visit 4 (5 - 7 Days after Tilmanocept Administration) The subject will report to the ACTRI research clinics for both Visits 3 and 4. These visits will include (see Table 1, Vital signs after at least 1 minute in a resting position (heart rate, blood pressure, and respiratory rate), Clinical Laboratory Evaluation: chemistry, hematology, Concomitant medication review, and Assessment and review of adverse events.

Blood and urine samples:

A total of 55 ml of blood and 30 ml of urine will be collected in this study. Samples will not be saved for future research. Genetic testing will not be done on any samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be required to satisfy the following criteria at the screening visit unless otherwise stated:

  1. The patient has provided written informed consent with HIPAA (Health Insurance Portability and Accountability Act) authorization before the initiation of any study-related procedures.
  2. The patient is at least 18 years of age at the time of consent.
  3. The patient has an ECOG performance status of Grade 0 - 2
  4. If of childbearing potential, the patient has a negative pregnancy test within 72 hours prior to administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year.
  5. Subjects will have a BMI of 18 to 49.9 kg/m2, inclusive, at screening.
  6. Meets clinical criteria described in the groups section above.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from the study.

  1. The patient is pregnant or lactating.
  2. The patient has participated in another investigational drug study within 3 months prior to Day 1.
  3. The subject has another significant medical condition requiring active surgical or medical intervention whose urgency would preclude participation in this study (active cardiac or pulmonary conditions,; ongoing ischemia or cardiac symptoms, uncorrected CAD or decompensated CHF).
  4. The subject has a Hemoglobin A1c>10.0
  5. The subject is on greater than 4 anti-hypertensives or has a a systolic blood pressure at time of screening greater than 160mm Hg.
  6. The patient has a suspected glomerulonephirtis, not including diabetic nephropathy, or hypertensive nephrosclerosis.
  7. The subject has a history of significant hypersensitivity, intolerance, or allergy to dextran or modified forms of dextran; unless approved by the Investigator.
  8. The subject has a history or presence of an acutely abnormal ECG, which, in the Investigator's opinion, is clinically significant.
  9. The subject has exceeded yearly radioactive dose of 30 mSv.
  10. The subject has a history of drug abuse or alcohol within 2 years before dose administration.
  11. The subjects used any prescription medications within 14 days prior to Day 1, except as allowed by the inclusion criteria or as deemed acceptable by the Investigator.
  12. The subject has poor peripheral venous access.
  13. The subject has donated blood within 30 days prior to Day 1, or plasma within 2 weeks prior to Day 1.
  14. The subject has received blood products within 2 months prior to Day 1.
  15. The subject has received any radiopharmaceutical within 7 days prior to the administration of Tc 99m tilmanocept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value in the kidney | Approximately 1 hour
  Time until 90% uptake in the kidney measured by SPECT/CT immediately after tilmanocept injection.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Hoh, MD, Principal Investigator — UC San Diego Medical Center
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Shared with an investigator on the supplemental award